CLINICAL TRIAL: NCT06840925
Title: A Phase 1, Randomized, Open-Label, 2-Way Crossover Clinical Trial in Healthy Participants to Evaluate the Relative Bioavailability of PRAX-628 Tablet Formulation Compared to Capsule Formulation
Brief Title: A Clinical Trial to Evaluate the Relative Bioavailability of PRAX-628
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Praxis Precision Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRAX-628-104
Record Dates: First submitted 2025-01-29; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Oral Dose 40mg PRAX-628 tablet then 4x10mg PRAX-628 capsules (Experimental): 40 mg PRAX-628 tablet followed by 4×10 mg PRAX-628 capsules administered orally.
  Interventions: Drug: PRAX-628
- Single Oral Dose 4x10mg PRAX-628 capsules then 40mg PRAX-628 tablet (Experimental): 4×10 mg PRAX-628 capsules followed by 40 mg PRAX-628 tablet administered orally.
  Interventions: Drug: PRAX-628

INTERVENTIONS:
Drug: PRAX-628 — Once daily oral

SUMMARY:
A phase I clinical trial to evaluate the relative bioavailability of PRAX-628 tablet formulation compared to capsule formulation

DETAILED DESCRIPTION:
This Phase 1, randomized, open-label, 2-way crossover clinical trial is designed to investigate the relative bioavailability, pharmacokinetics (PK), safety, and tolerability of PRAX628 tablet formulation and PRAX-628 capsule formulation in healthy male or female participants.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 50 kg with body mass index (BMI) between 18 and 32 kg/m2
* Is in good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations
* All females have a negative pregnancy test and are not planning to get pregnant for the duration of the trial
* Female of non-childbearing potential by reason of surgery or at least 1 year post menopause
* Additional inclusion criteria apply and will be assessed by the study team

Exclusion Criteria:

* Any clinically significant abnormalities, medical, or psychiatric conditions identified by a detailed medical history, or physical examination
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs. Examples of such conditions include (but are not limited to):

  1. History of inflammatory bowel syndrome, gastritis, gastrointestinal or rectal bleeding
  2. History of major gastrointestinal tract surgery (ie, gastrectomy, bowel resection, cholecystectomy etc.)
  3. History or evidence of pancreatic injury or pancreatitis
* History or presence of impaired renal function supported by estimated glomerular filtration rate [eGFR]<60 mL/min/1.73m2 or clinically significant abnormal urinary constituents (eg, protein)
* History of cancer except for nonmelanoma skin cancer resected >2 years ago and that has been definitively treated and considered cured.
* History of any lifetime suicide attempt or active suicidal ideation with intent as indicated by a "Yes" response to either Question 4 or 5 on the C-SSRS "Baseline/ Screening" version
* History of left bundle branch block, arrhythmias, Brugada syndrome, congenital heart disease, familial short QT syndrome, or family (first degree relative) history of sudden death, ventricular or clinically significant arrhythmias, including idiopathic ventricular fibrillation.
* Abnormal standard 12-lead ECG after at least 5 minutes resting in the supine position
* Abnormal vital signs after at least 5 minutes resting in the supine position:
* Has any of the following: a serum total bilirubin value >1.1× the upper limit of normal (ULN), a serum alanine aminotransferase (ALT) value >1.5×ULN, or aspartate aminotransferase (AST) value >1.5×ULN
* Serology test positive for human immunodeficiency virus (HIV), or hepatitis B or C
* Known allergy or hypersensitivity to any component of the formulation of PRAX 628 or history of severe allergy or anaphylaxis to a drug, food, or other exposure
* Use of any experimental or investigational drug or device within 30 days prior to the first dose of study drug or 5 times the terminal half-life of the drug, whichever is longer
* Use of systemic prescription medications; or over-the-counter medication, including multivitamins; and dietary and herbal supplements within 2 weeks or 5 times the terminal half-life of the medication prior to the first dose of study drug (whichever is longer) and for the duration of the trial
* Donation of blood within 1 month prior to Screening, plasma within 1 week prior to Screening, or platelets within 6 weeks prior to Screening
* Any vaccination within 28 days of the first dose of study drug
* Additional exclusion criteria apply and will be assessed by the study team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the relative bioavailability of single 40 mg oral doses of PRAX-628 tablet as compared to PRAX-628 capsules | 28 days
  Geometric mean ratio (90% CI) for maximum observed plasma concentration (Cmax)
To assess the relative bioavailability of single 40 mg oral doses of PRAX-628 tablet as compared to PRAX-628 capsules | 28 days
  Area under the plasma concentration time curve from time zero to infinity (AUCinf) of a single dose of PRAX-628 40 mg tablet (test), and the same dose delivered with PRAX-628 10 mg capsules (reference)

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 28 days
  Plasma concentrations of PRAX-628 (Cmax)
To evaluate the pharmacokinetics (PK) of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 28 days
  Time to maximum plasma drug concentration (tmax)
To evaluate the pharmacokinetics (PK) of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 28 days
  Area under the plasma concentration versus time curve (AUC)
To evaluate the safety and tolerability of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 32 days
  Incidence and severity of adverse events (AEs)
To evaluate the safety and tolerability of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 32 days
  Change in tympanic temperature in Celsius
To evaluate the safety and tolerability of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 32 days
  Change in heart rate in beats per minute
To evaluate the safety and tolerability of single 40 mg oral doses of PRAX-628 tablet and PRAX-628 capsules | 32 days
  Change in blood pressure in mm/Hg
To evaluate the safety and tolerability of single 40 mg oral doses of PRAX-628 tablet and PRAX 628 capsules | 32 days
  Change in respiratory rate in breaths per minute
Number of Participants With Clinically Significant Changes in Chemistry parameters | 32 days
  The principal investigator (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.
Number of Participants With Clinically Significant Changes in Hematology parameters | 32 days
  The principal investigator (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.
Number of Participants With Clinically Significant Changes in Urinalysis | 32 days
  The Princpal investigatort (PI) or sub investigator will review the laboratory report and document this review. Any clinically significant adverse changes occurring during the clinical trial will be documented as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Development, Study Director — Praxis Precision Medicines
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia